CLINICAL TRIAL: NCT04920630
Title: TRAIN Your Sleep: Treating Adolescent Insomnia With Cognitive Behavioral Therapy for Insomnia (CBT-I)
Brief Title: TRAIN Your Sleep; Treating Adolescent Insomnia With Cognitive Behavioral Therapy for Insomnia (CBT-I)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research team members no longer employed. Determination made to utilize pilot data already obtained and close study to enrollment.
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Amy E. Williams, Associate Professor of Clinical Psychiatry, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009842860
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Insomnia; Chronic Pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-I (Experimental): 5-weekly Cognitive Behavioral Therapy for Insomnia group therapy sessions conducted virtually.
  Interventions: Behavioral: Cognitive Behavioral Therapy - Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy - Insomnia (CBT-I) — CBT-I will be delivered via 5 weekly virtual group therapy sessions. Session content is manualized and adapted from existing CBT-I protocols to be relevant to a virtual adolescent group and will include: Session 1 - Introduction of group members, group rules, psychoeducation regarding sleep, and instructions on completion of sleep log. Session 2 - Review sleep log, sleep hygiene, relaxation training, and stimulus control. Session 3 - Review sleep log, sleep restriction, and cognitive strategies (positive self-statements, worry management). Session 4 - Review sleep log and sleep restriction, and problem-solving barriers. Session 5 - Maintenance and relapse prevention.
  Other Names: CBT-I

SUMMARY:
The primary aim of this study is to understand how insomnia contributes to chronic pain in youth. Specifically, the investigators are interested in how insomnia and the treatment of insomnia impact emotional states and the body's ability to efficiently modulate pain, either to increase or decrease pain perception. It is hypothesized that insomnia is associated with increased negative emotional states and impaired pain modulation, which will improve after treatment of insomnia. In this project, the objectives are to 1) evaluate the role of pain modulation as a potential mechanism through which insomnia impacts pain symptoms, and 2) evaluate the role of negative affect as mediators of the impact of insomnia on pain modulation.

Study participation will consist of a baseline assessment, a 5 session (once per week) virtual group cognitive behavioral therapy for insomnia (CBT-I) intervention, and a follow-up assessment. Investigators will also ask teen participants to complete the consensus sleep diary daily for 7 days prior to the baseline and follow up study visits. Assessment visits will consist of two types of assessments, questionnaires and quantitative sensory testing (QST). Participating parents and teens will complete questionnaires (both child and parent report) assessing the child's pain, sleep, and psycho-social variables. QST will assess pain inhibition via conditioned pain modulation (CPM) and pain facilitation via temporal summation (TS).

ELIGIBILITY:
Youth Inclusion Criteria:

* Aged 12 to 17 years.
* Meets criteria for insomnia with or without comorbid chronic musculoskeletal pain.
* Parent/guardian available to provide consent.
* Patient and a primary caregiver are able to independently read and understand English well enough to provide informed consent and complete study procedures.
* Access to email, internet, and audio and video call capabilities.

Parent/Guardian Inclusion Criteria:

* Parent/legal guardian of a child meeting above eligibility criteria
* Able to independently read and understand English well enough to provide informed consent and complete study questionnaires.

Youth Exclusion Criteria:

* History of cardiac or neuromuscular disorder
* Parent-report of child's use of Opioid medications (i.e., fentanyl, morphine, hydromorphone, methadone, hydrocodone, oxycodone) that cannot be discontinued for 7 days prior to study visits.
* Inadequate proficiency in English or a developmental disability that interferes with informed consent/assent or completion of study procedures.
* History of obstructive sleep apnea, restless leg syndrome, or narcolepsy.
* History of bipolar disorder and/or manic episodes
* Diagnosis of epilepsy.
* Currently in foster care or considered a ward of the state.
* History of Raynaud Syndrome.
* Active suicidal ideation, intent or plan in the past month.

Parent Exclusion Criteria:

• Inadequate proficiency in English or a developmental disability that interferes with informed consent or completion of questionnaires.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Conditioned Pain Modulation (CPM) | 1-4 weeks post-treatment
  Heat pain threshold (test stimulus) will be assessed on the volar surface of the dominant forearm twice before before, during, and after immersion (for 1 minute) of the non-dominant hand in a circulated cold-water bath (conditioning stimulus) maintained at 5˚C ±1˚C. Heat pain threshold will be assessed via the method of limits. Subjects will be instructed to push a button as soon as the heat feels painful, which will stop the trial. Immediately before and after the CPM assessment, the subjects' non-dominant hand will be placed in a room-temperature water bath (20-25˚C) for 2 minutes. The CPM effect will be calculated as a difference score: heat pain threshold during conditioning stimulus minus baseline. A negative score indicates pain inhibition.
Change from baseline Temporal Summation of Pain (TS) | 1-4 weeks post-treatment
  Temporal summation will be assessed via a series of 10 brief (~0.5s duration for peak, total time for heating, peak, and cooling <1.5s) heat pulses (48˚C) delivered via a Medoc Thermal Sensory Analyzer-2 thermode positioned on the volar surface of the forearm. Time between each peak will be 3 seconds. Subjects will provide a verbal pain rating immediately after the first and last heat pulse is delivered. Pain ratings will be made on a 0-100 numerical rating scale (0=no pain, 100=most pain imaginable), which will be displayed during the assessment. Temporal summation will be calculated as a difference score (i.e., pain during final stimulus minus pain during initial stimulus), with a positive score indicating pain facilitation due to temporal summation.

SECONDARY OUTCOMES:
Change from baseline score on Generalized Anxiety Disorder -7 | 1-4 weeks post-treatment
  Generalized Anxiety Disorder - 7 (GAD-7). The GAD-7 is a 7 item screener for anxiety focused on symptoms of anxiety over the past week. Each item is scores on a 0-3 scale and summed to create a total score that ranges from 0-21.
Change from baseline score on Patient Health Questionnaire - 9 Adolescent Form (PHQ9-A). | 1-4 weeks post-treatment
  The PHQ9-A is a validated 9 item self-report scale (4-point Likert scale) assessing symptoms of depression. Scores range from 0-27 with 0-4 indicating no or minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.
Change from Baseline Score on Positive and Negative Affect Schedule (PANAS) | 1-4 weeks post-treatment
  he PANAS is a 20-item self- and parent-report measure assessing positive and negative affect. Responses are made on a 5-point Likert scale. A separate score is calculated for negative (10 items) and positive (10 items) affect and higher scores reflect higher levels of experienced affect.
Change from baseline score on Pediatric Insomnia Severity Index (PISI) | 1-4 weeks post-treatment
  The PISI is a 6-item parent- and child-report scale measuring insomnia severity. Total scores range from 0-30 with higher scores reflecting greater insomnia severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Childre, Indianapolis, Indiana, United States